CLINICAL TRIAL: NCT05412342
Title: Observational Study to Characterize the Relationship Between Preoperative Depressive Symptoms and Opioid Use/Misuse After Surgery
Brief Title: Characterizing the Association Between Preoperative Depressive Symptoms and Opioid Use/Misuse After Surgery
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jennifer Hah, Assistant Professor, Stanford University
Other Study IDs: 43163
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Opioid Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing elective operations: We will follow a prospective cohort of 558 patients, undergoing any elective surgery at Stanford Hospital. Subjects will undergo baseline and longitudinal testing via a (including NIH Patient-Reported Outcomes Measurement Information System- PROMIS measures of emotional distress). After surgery, participants will report weekly changes in opioid use, pain, and adverse events; and monthly changes in opioid misuse for 1 year.

SUMMARY:
This observational study aims to characterize the relationship between preoperative depressive symptoms and opioid use/ misuse after surgery using a perioperative learning health care system. We will follow a prospective cohort of patients undergoing elective surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18+
2. Planning to undergo surgery
3. English speaking
4. Ability and willingness to complete questionnaires and assessments

Exclusion Criteria:

1. Any conditions causing inability to complete assessments (education, cognitive ability, mental status, medical status)
2. Known Pregnancy
3. Elevated Suicidality
4. Enrollment in a conflicting perioperative trial

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgery at Stanford Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 718 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2024-03-03 (Actual); Study Completion 2024-03-03 (Actual)

PRIMARY OUTCOMES:
Time to Opioid Cessation | Assessed after surgery up to 1 year

SECONDARY OUTCOMES:
Opioid Misuse | Assessed after surgery up to 1 year
  Participant score on the Current Opioid Misuse Measure will be used to assess opioid misuse

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Palo Alto, California
  - Stanford Health Care, Stanford, California

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT05412342/ICF_000.pdf